CLINICAL TRIAL: NCT01519258
Title: Performance of NAVA as Lung Protective Mechanical Ventilation in Patients With Acute Respiratory Distress Syndrome
Brief Title: Mechanical Ventilation With Neurally-Adjusted Ventilatory Assist in Patients With ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011/20225-1 FAPESP
Record Dates: First submitted 2011-12-07; First posted 2012-01-26 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSV (Active Comparator): Patients will be ventilated with the a conventional mode of ventilation called Pressure Support Ventilation (PSV) for 15 minutes. Mechanical ventilator settings will be set to match the tidal volume applied by the ICU team, in accordance to current standard of care recommendations.
  Interventions: Other: Pressure Support ventilation
- NAVA (Experimental): Patients will be ventilated with NAVA for 15 minutes. Nava level will be titrated prior to randomization, to deliver the same peak of airway pressure obtained with the active comparator, PSV. The resulting tidal volume should match the tidal volume applied by the ICU team, in accordance to current standard of care recommendations.
  Interventions: Device: NAVA

INTERVENTIONS:
Other: Pressure Support ventilation — Patients will receive usual care during the period of ventilation on the Pressure Support. The same ventilator, the Servoi (maquet, Sweden) will be used.
  Arms: PSV
Device: NAVA — Patients will be ventilated with NAVA for 15 minutes. Back up settings in pressure support mode will be set in case the esophageal catheter is misplaced, and back up settings in pressure control ventilation will be set in case no inspiratory efforts are detected for longer than 15 seconds
  Arms: NAVA

SUMMARY:
Neurally-Adjusted Ventilatory Assist (NAVA) is a ventilatory mode that uses the electrical activity of the diaphragm to control the mechanical ventilator, offering inspiratory assistance in proportion to respiratory effort to patients who need artificial ventilatory support. It has been shown to improve the interaction between the patient and the mechanical ventilator in several clinical situations, but no previous studies have tried to use it for patients with a severe type of respiratory insufficiency, called Acute Respiratory Distress Syndrome (ARDS). Patients with ARDS benefit from a mechanical ventilatory strategy that includes low inspiratory volumes (tidal volumes) and limited airway pressures, but the application of such strategy frequently requires high levels of sedation. The investigators' hypothesis is that NAVA can be used for patients with ARDS, and that it will not be associated with excessive tidal volumes or elevated airway pressures.

DETAILED DESCRIPTION:
Neurally Adjusted ventilatory-Assist(NAVA) is an assisted ventilatory mode that captures the electrical activity of the diaphragm and uses it to initiate and terminate the inspiratory phase, offering inspiratory assistance in proportion to patient effort, cycle by cycle. Studies in animals and humans have shown that NAVA reduces the work of breathing and improves patient-ventilator interaction in comparison with traditional modes. Because it is an assisted mode, its use requires less sedation.

The use of NAVA could contribute to the reduction of complications of prolonged mechanical ventilation in patients with Acute Respiratory Distress Syndrome (ARDS) submitted to protective ventilation with low tidal volumes and limited plateau pressure. However, there are no studies with NAVA in the acute phase of ARDS, in which assisted-controlled modes are generally used, allowing for adjustment of tidal volume and/or plateau pressure.

With this project, the investigators intend to evaluate the behavior of NAVA mode in the acute phase of mechanical ventilation in ARDS patients, to assess whether this mode can be used to deliver an assisted lung protective ventilation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation for more than 24 hours;
* Diagnosis of ARDS
* Clinical indication of lung protective mechanical ventilation by the ICU team;
* Presence of active inspiratory efforts for more than 6 hours

Exclusion Criteria:

* Patients under 18 years;
* Pregnant women;
* Trauma or burns of the face that hinder the passage of gastro-esophageal catheter;
* Nasal pathologies that prevent the progression of gastro-esophageal catheter;
* Ulcers of the esophagus or stomach;
* Documented esophageal varices;
* Tracheostomized patients;
* Instability of the chest wall or diaphragmatic injury;
* Hemodynamic instability, defined as the need to increase vasoactive drugs in the last two hours in order to maintain the mean arterial pressure above 60 mmHg).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Tidal volume | 15 min
  Tidal volume will be recorded breath by breath for 15 minutes

SECONDARY OUTCOMES:
respiratory rate | 15 min
  Respiratory rate will be recorded breath by breath for 15 minutes
Prolonged NAVA ventilation | 3 hours
  patients will be kept on NAVA for three hours after the first part of the protocol, to evaluate the feasibility of ventilating these patients with NAVA for prolonged periods

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Ferreira, M.D., Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Diniz-Silva F, Moriya HT, Alencar AM, Amato MBP, Carvalho CRR, Ferreira JC. Neurally adjusted ventilatory assist vs. pressure support to deliver protective mechanical ventilation in patients with acute respiratory distress syndrome: a randomized crossover trial. Ann Intensive Care. 2020 Feb 10;10(1):18. doi: 10.1186/s13613-020-0638-0. PMID 32040785